CLINICAL TRIAL: NCT06313879
Title: The Effect of Tele-Education Provided to Parents of Children With Hydrocephalus and Ventriculoperitoneal Shunt on Their Anxiety and Self-Efficacy
Brief Title: The Effect of Education Given to Parents of Children With Ventriculoperitoneal Shunt on Their Anxiety and Self-efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Sevinc Aka, Principal Investigator, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PamukkaleU-SBE-SA-01
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hydrocephalus in Children
Keywords: online education; ventriculoperitoneal shunt; hydrocephalus in children; self sufficiency; parental anxiety

STUDY DESIGN:
Intervention Model Description: Two groups: comparative experiment and control
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trained parent group (Experimental): The experimental group will be given a total of 6 hours of training for 2 weeks, and they will be asked to fill out the State and Trait Anxiety Scale and the General Self-Efficacy Scale before and after the training. After 3 months of counseling, the scales will be filled in again.
  Interventions: Behavioral: Tele-education and Counseling Program
- uneducated parent group (No Intervention): The control group will be asked to fill out the State and Trait Anxiety Scale and the General Self-Efficacy Scale at the first interview. After 2 weeks, they will be asked to fill out the scales simultaneously with the experimental group, without any training. They will be asked to fill out the Parental Knowledge Test, State and Trait Anxiety Scale, and General Self-Efficacy Scale simultaneously with the experimental group, without any intervention for 3 months.

INTERVENTIONS:
Behavioral: Tele-education and Counseling Program — A structured online behavioral program that provides video-based education and scheduled tele-counseling sessions for parents of children with ventriculoperitoneal (VP) shunts. The intervention includes educational modules, digital informational materials, and tele-counseling follow-ups delivered over a 3-month period.
  Arms: trained parent group

SUMMARY:
This study aims to evaluate the effect of tele-education given to parents of children with ventriculoperitoneal shunt on their anxiety and self-efficacy.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of tele-education given to parents of children with ventriculoperitoneal shunt on their anxiety and self-efficacy. The type of research was planned as a prospective, randomized controlled experimental study with a pretest-posttest control group. The research will be conducted online with the parents of children with ventriküloperitoneal shunts at Pamukkale University Hospital. The data of the research will be collected between March 2024 and February 2025. In data collection, a personal information form will be used to determine the socio-demographic characteristics of the participants, a parent knowledge test will be used to evaluate their knowledge levels, and the General Self-Efficacy Scale and State and Trait Anxiety Scale will be used to evaluate the dependent variables. It was determined that 60 parents should participate in the study, 30 for the experimental group and 30 for the control group. As the randomization method, "simple randomization" will be used to ensure an equal number of samples in the experimental and control groups. Randomization will be done using the www.randomizer.org application. The data will be analyzed with the SPSS (23.0) package program. Continuous variables will be given as mean ± standard deviation and categorical variables will be given as number and percentage. Significance Test of Difference Between Two Means in comparing independent group differences when parametric test assumptions are met; When parametric test assumptions are not met, Mann-Whitney U test will be used to compare independent group differences.

ELIGIBILITY:
Inclusion Criteria:

Parent of a child aged 0-6 years with a VP shunt Able to access the internet Willing to participate Able to complete online questionnaires

Exclusion Criteria:

Difficulty accessing the internet Not participating in the online group Not responding to questionnaires Having a child older than 6 years with a VP shunt

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
State and Trait Anxiety Scale | Two months
  This inventory includes the State and Trait Anxiety Scales. Each contains 20 items. In State Anxiety, the options "Never", "Somewhat", "A lot", "Completely" are used, and in Trait Anxiety the options "Almost Never", "Sometimes", "Most of the Time", "Almost Always" are used. Weights of 1 in positive expressions are converted to 4, and weights of 4 in negative expressions are converted to 1. Certain items have reverse expressions and scoring is done accordingly. 10 items in State Anxiety and 7 items in Trait Anxiety contain reverse wording. For scoring, the scores of the reverse expressions are subtracted from the direct scores and fixed values (50 points for the state anxiety scale, 35 points for the trait anxiety scale) are added. The total score on both scales is between 20-80. A high score indicates high anxiety, a low score indicates low anxiety.

SECONDARY OUTCOMES:
General Self-Efficacy Scale | Two months
  The scale was created using a five-point Likert-type scale from 1 to 5 (1 = Not at all; 5 = Very Good) and contains 17 items in total. Items 2, 4, 5, 6, 7, 10, 11, 12, 14, 16 and 17 in the scale are evaluated by reverse scoring method. The research examines self-efficacy in terms of initiation (items 2, 4, 5, 6, 7, 10, 11, 12 and 17), resistance (items 3, 13, 14, 15 and 16) and maintenance effort-persistence (items 1, 16). It is analyzed in three different sub-dimensions: items 8 and 9).

CONTACTS AND LOCATIONS:
Overall Officials: Türkan Turan Professor Doctor, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University Hospital, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No